CLINICAL TRIAL: NCT03317639
Title: Improving In-hospital Stroke Service Utilisation (MISSION) in China: A Cluster Randomised Trial of Interventions to Shorten Door to Needle Times
Brief Title: Improving In-hospital Stroke Service Utilisation in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shaoxing Second Hospital (Other); Haining People' s Hospital (Unknown); Haiyan People' s Hospital (Unknown); Huzhou No.1 People' s Hospital (Unknown); Jiashan No.1 People' s Hospital (Unknown); Ningbo Medical Center Lihuili Hospital (Other Government); Tongxiang No.1 People' s Hospital (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); Yiwu Central Hospital (Other); Yongkang No.1 People' s Hospital (Unknown); Yuyao People's Hospital (Other); Deqing People' s Hospital (Unknown); Dongyang People's Hospital (Other); Jinhua People' s Hospital (Unknown); Lishui People' s Hospital (Unknown); Lin' an People' s Hospital (Unknown); Longquan People' s Hospital (Unknown); Qingtian People' s Hospital (Unknown); Shaoxing Central Hospital (Other); Wenzhou Central Hospital (Other); Xiangshan No.1 People' s Hospital (Unknown); The Central Hospital of Lishui City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MISSION CHINA
Record Dates: First submitted 2017-10-15; First posted 2017-10-23 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-01

CONDITIONS: Thrombolytic Therapy; Acute Stroke; Door to Treatment Time; Quality Improvement
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- an intervention arm (Experimental): Hospitals in the intervention arm will receive a multi-components intervention based on the Behaviour Change Wheel model
  Interventions: Behavioral: Behaviour Change Wheel model guided intervention
- a control arm (No Intervention): hospitals in the control arm will receive no intervention and maintain existing care

INTERVENTIONS:
Behavioral: Behaviour Change Wheel model guided intervention — Interventions are developed on a psychological model, the Behaviour Change Wheel (BCW) .The fundamental of BCW consists of three essential elements: capability, motivation, and opportunity. Improving individual's capability, providing motivation, and increasing opportunities are goals of behaviour change intervention. To achieve the goals, 9 intervention components have been proposed in the BCW framework, and 6 components will be used in current study.
  Arms: an intervention arm

SUMMARY:
A cluster randomised controlled trial will be conducted, using hospital as randomisation unit. Hospitals in Zhejiang Province, China, will be randomised into two arms (1:1): an intervention arm and a control arm. Hospitals in the intervention arm will receive a multi-components intervention based on the Behaviour Change Wheel model, whereas hospitals in the control arm will receive no intervention and maintain existing care. The randomisation will be conducted after one-year baseline data collection. The following baseline data will be used for randomisation match: hospital classification, beds in stroke centre, thrombolysis patient number, and percentage of patients receiving thrombolysis within 60 minutes of stroke onset. Hospitals with no stroke centre or with <20 cases received thrombolysis per year will be excluded from the study. The primary outcome will be difference between intervention arm and control arm in the percentage of patients receiving thrombolysis within 60 minutes of stroke onset on the follow-up stage (post-intervention).

ELIGIBILITY:
Inclusion Criteria:

* AIS patients receiving IVT within 4.5 hours

Exclusion Criteria:

* Patients who are not willing to attend this trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1634 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Difference in the percentage of patients who Door-to-Needle Time≤60min | Up to 24 hours
  Difference between intervention arm and control arm in the percentage of patients receiving thrombolysis within 60 minutes of stroke onset on the follow-up stage

SECONDARY OUTCOMES:
Door-to-needle time | Up to 24 hours
  The time between hospital arrival and the initiation of IVT
Onset-to-needle time | Up to 24 hours
  The time between the symptom onset and the initiation of IVT
modified Rankin Scale score at discharge | Up to 3 month
  modified Rankin Scale score at discharge, on which scores range from 0 (no neurologic deficit) to 6 (death)
Symptomatic intracranial hemorrhage | At 24 hours
  Intracranial hemorrhage at 24 hours associated with an increase of ≥4 points of NIHSS score from baseline, according to European Cooperative Acute Stroke Study (ECASS) II trial
Favorable neurological outcomes | At 90 days
  Score of 0 to 1 on the modified Rankin Scale, on which scores range from 0 (no neurologic deficit) to 6 (death)
Death | Up to 3 month
  Death at discharge

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Lynch EA, Bulto LN, Cheng H, Craig L, Luker JA, Bagot KL, Thayabaranathan T, Janssen H, McInnes E, Middleton S, Cadilhac DA. Interventions for the uptake of evidence-based recommendations in acute stroke settings. Cochrane Database Syst Rev. 2023 Aug 11;8(8):CD012520. doi: 10.1002/14651858.CD012520.pub2. PMID 37565934
- [Derived] Zhong W, Lin L, Gong X, Chen Z, Chen Y, Yan S, Zhou Y, Zhang X, Hu H, Tong L, Cheng C, Gu Q, Chen Y, Yu X, Huang Y, Yuan C, Lou M; MISSION investigators. Evaluation of a multicomponent intervention to shorten thrombolytic door-to-needle time in stroke patients in China (MISSION): A cluster-randomized controlled trial. PLoS Med. 2022 Jul 5;19(7):e1004034. doi: 10.1371/journal.pmed.1004034. eCollection 2022 Jul. PMID 35788767
- [Derived] Wang J, Gong X, Zhong W, Zhou Y, Lou M. Novel Prehospital Triage Scale for Detecting Large Vessel Occlusion and Its Cause. J Am Heart Assoc. 2021 Sep 7;10(17):e021201. doi: 10.1161/JAHA.121.021201. Epub 2021 Aug 21. PMID 34423654